CLINICAL TRIAL: NCT05878691
Title: A Phase 1, Open Label First In Human Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HPK1 Inhibitor GRC 54276 Alone and in Combination With Anti-PD-1 Monoclonal Antibody Pembrolizumab or Anti-PD-L1 Atezolizumab in Subjects With Advanced Solid Tumors and Lymphomas.
Brief Title: A Study of GRC 54276 in Participants With Advanced Solid Tumors and Lymphomas.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GRC 54276-101; CTRI/2022/05/042484 (Registry Identifier: Clinical Trials Registry-India)
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor; Lymphoma
Keywords: Solid tumor; Lymphoma; MTD
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GRC 54276 (Experimental)
  Interventions: Drug: GRC 54276
- GRC 54276 with pembrolizumab (Experimental)
  Interventions: Drug: GRC 54276 + Pembrolizumab
- GRC 54276 with atezolizumab (Experimental)
  Interventions: Drug: GRC 54276 + Atezolizumab

INTERVENTIONS:
Drug: GRC 54276 — Part 1a: GRC 54276 QD will be administered orally from Day 1 to Day 21 in a 21-day treatment cycle.
  Part 2: GRC 54276 monotherapy therapy will commence after establishment of the MTD and/or RP2D for monotherapy arm.
  Arms: GRC 54276
Drug: GRC 54276 + Pembrolizumab — Part 1b: GRC 54276 QD will be administered orally in combination with fixed dose of pembrolizumab IV every 21 days.
  Part 2: GRC 54276 in combination with pembrolizumab will commence after establishment of the MTD and/or RP2D for combination therapy arm.
  Arms: GRC 54276 with pembrolizumab
Drug: GRC 54276 + Atezolizumab — Part 1b: GRC 54276 QD will be administered orally in combination with fixed dose of atezolizumab IV every 21 days.
  Part 2: GRC 54276 in combination with atezolizumab will commence after establishment of the MTD and/or RP2D for combination therapy arm.
  Arms: GRC 54276 with atezolizumab

SUMMARY:
This is first in human (FIH) study to a) evaluate the safety and tolerability profile of GRC54276, b) determine the maximum tolerated dose (MTD) and recommended Phase 2 doses (RP2D), and c) pharmacokinetic profile of GRC54276 alone and in combination with pembrolizumab or atezolizumab in participants with advanced solid tumors and lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (≥18 years of age) with histologically or cytologically confirmed advanced, metastatic, unresectable solid tumors or lymphomas who have previously received standard systemic therapy or for whom treatment is not accessible, not tolerated or refused, have progressed after ≥1 of systemic therapies for recurrent/metastatic disease and who have not received prior therapy targeting HPK1.
2. At least 1 measurable lesion as defined per RECIST 1.1. The target lesion(s) selected have not been previously treated with local therapy or the target lesion(s) selected that are within the field of prior local therapy have subsequently progressed as defined by RECIST 1.1.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1 measured within 72 hours of treatment.
4. Predicted life expectancy of ≥3 months.
5. Adequate organ function as indicated by the following laboratory values up to first dose of study drug: Hemoglobin ≥9.0 g/dL, Absolute neutrophil count ≥1.5 x 109/L, Serum total bilirubin ≤1.5 x ULN (<3 x ULN for participants with Gilbert syndrome), AST and ALT ≤2.5 x ULN (≤5 x ULNs for participants with hepatocellular carcinoma or liver metastases).
6. Adequate renal function as indicated by creatinine clearance of ≥60mL/min calculated using Cokroft-Gault method.
7. Adequate cardiac function, left ventricular ejection fraction (LVEF) of ≥50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO).
8. For Part 2, dose expansion cohorts inclusion criteria specific to tumor types will be updated after completion of Part 1.

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study drug or interpretation of subject safety or study results.
2. Subjects with uncontrolled or untreated brain metastasis or leptomeningeal disease. Subjects with equivocal findings or with confirmed brain metastases are eligible provided that they are asymptomatic and radiologically stable without the need for corticosteroid treatment for at least 4 weeks prior to the first dose of study drug(s)
3. Any active malignancy ≤2 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast)
4. Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before the first dose of study drug(s), with the following exceptions:

   1. Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
5. Pregnant/planning to be pregnant or breast-feeding women.
6. Any important medical illness or abnormal laboratory finding that would increase the risk of participating in this study (based on the investigator's judgment).
7. Any known severe allergic reaction to pembrolizumab/atezolizumab or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities to establish the maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | 18 weeks
  Percentage of participants with dose limiting toxicities associated with GRC54276 alone or GRC54276 combined with pembrolizumab or atezolizumab during the first cycle. Toxicity will be assessed using the NCI CTCAE Version 5.0.
Incidence of treatment-emergent adverse events and serious adverse events | up to 120 days
  Percentage of participants who experience treatment-emergent adverse events and serious adverse events when given GRC54276 as a single agent and in combination with pembrolizumab or atezolizumab.
Changes in the laboratory safety values from baseline to end of safety follow-up | up to 120 days
  Percentage of participants who experience changes in the laboratory safety values when given GRC54276 as a single agent and in combination with pembrolizumab or atezolizumab.
Pharmacokinetic profile of GRC54276- Maximum plasma concentration (Cmax) | up to 22 days
  The maximum measured plasma concentration after single or multiple dosing, tabulated by dose group and day of dosing.
Pharmacokinetic profile of GRC54276- Time to Cmax (Tmax) | up to 22 days
  The time to achieve Cmax after single or multiple dosing, tabulated by dose group and day of dosing.
Pharmacokinetic profile of GRC54276- Area under the curve (AUC) | up to 22 days
  Area under plasma concentration versus time curve from time 0 to time of least measurable concentration or the dosing interval, tabulated by dose group and day of dosing.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 9 months
  Proportion of participants with a best response of complete response or partial response best on RECIST 1.1.
Best overall response rate | up to 9 months
  Complete response, partial response, stable disease, and progressive disease, evaluated according to RECIST 1.1.
Disease control rate | up to 9 months
  The percentage of participants who have achieved stable disease or complete response or partial response according to RECIST 1.1. for the entire duration of the study.
Duration of response | up to 9 months
  The time from first documentation of complete response or partial response to the first documentation of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Gupta, Study Director — Glenmark Pharmaceuticals Ltd.
Locations (18):
- United States (2):
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Froedtert & Medical College of Wisconsin - Froedtert Hospital - Clinical Cancer Center, Milwaukee, Wisconsin
- India (16):
  - Hcg City Cancer Centre, Vijayawada, Andhra Pradesh
  - Mahatma Gandhi Cancer Hospital and Research Institute, Visakhapatnam, Andhra Pradesh
  - Artemis Hospital, Gurgaon, Haryana
  - Health Care Global Enterprises Ltd (HCG), Bangalore, Karnataka
  - Vydehi Hospital, Bangalore, Karnataka
  - Cytecare Hospitals Pvt Ltd., Bengaluru, Karnataka
  - Aster CMI Hospital, Bengaluru, Karnataka
  - Malabar Cancer Centre, Kannur, Kerala
  - Krupamayi Hospitals, Aurangabad, Maharashtra
  - PD Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Sankalp Hospital, Nashik, Maharashtra
  - Bhaktivedanta Hospital and Research Institute, Thane, Maharashtra
  - AIG Hospitals, (A unit of asian Institute of Gastroenterology), Hyderabad, Telangana
  - Basavatarakam Indo American Cancer Hospital Research Institute, Hyderabad, Telangana
  - Max Superspeciality Hospital, Delhi